CLINICAL TRIAL: NCT06360445
Title: A Randomized, Open-Label, 2-formulation, Single-Dose, 2-Period Crossover Bioequivalence Study of Olaparib Tablets Under Fasting and Fed Conditions in Healthy Subjects
Brief Title: Bioequivalence Study of Olaparib Tablets Under Fasting and Fed Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD1912BE202201
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: 2-period Crossover Assignment
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Olaparib Tablet test formulation 100mg (Experimental): Treatment A: During the study session, healthy subjects were administered a single dose of Olaparib Tablet test formulation100mg under Fasting conditions(test)
  Interventions: Drug: Olaparib Tablet test formulation 100mg
- Olaparib Tablet reference formulation 100mg (Active Comparator): Treatment B: During the study session, healthy subjects were administered a single dose of Olaparib Tablet reference formulation 100mg under Fasting conditions(reference for Treatment A)
  Interventions: Drug: Olaparib Tablet reference formulation 100mg
- Olaparib Tablet test formulation 150mg(fast) (Experimental): Treatment C: During the study session, healthy subjects were administered a single dose of Olaparib Tablet test formulation 150mg under Fasting conditions(test)
  Interventions: Drug: Olaparib Tablet test formulation 150mg
- Olaparib Tablet reference formulation 150mg(fast) (Active Comparator): Treatment D: During the study session, healthy subjects were administered a single dose of Olaparib Tablet reference formulation 150mg under Fasting conditions(reference for Treatment C)
  Interventions: Drug: Olaparib Tablet reference formulation 150mg
- Olaparib Tablet test formulation 150mg(fed) (Experimental): Treatment E: During the study session, healthy subjects were administered a single dose of Olaparib Tablet test formulation 150mg under Fed conditions(test)
  Interventions: Drug: Olaparib Tablet test formulation 150mg
- Olaparib Tablet reference formulation 150mg(fed) (Active Comparator): Treatment F: During the study session, healthy subjects were administered a single dose of Olaparib Tablet reference formulation 150mg under Fed conditions(reference for Treatment E)
  Interventions: Drug: Olaparib Tablet reference formulation 150mg

INTERVENTIONS:
Drug: Olaparib Tablet test formulation 100mg — A generic product manufactured by CSPC Ouyi Pharmaceutical Co., Ltd.
  Arms: Olaparib Tablet test formulation 100mg
Drug: Olaparib Tablet reference formulation 100mg — Olaparib Tablet reference formulation 100mg were used as a comparator drug for the bioequivalence study, manufactured by AbbVie Limited.
  Arms: Olaparib Tablet reference formulation 100mg
Drug: Olaparib Tablet test formulation 150mg — Olaparib Tablet reference formulation 150mg were used as a comparator drug for the bioequivalence study, manufactured by AbbVie Limited.
  Arms: Olaparib Tablet test formulation 150mg(fast); Olaparib Tablet test formulation 150mg(fed)
Drug: Olaparib Tablet reference formulation 150mg — Olaparib Tablet reference formulation 150mg were used as a comparator drug for the bioequivalence study, manufactured by AbbVie Limited.
  Arms: Olaparib Tablet reference formulation 150mg(fast); Olaparib Tablet reference formulation 150mg(fed)

SUMMARY:
This Study is a Randomized, Open-Label, 2-formulation, Single-Dose, 2-Period Crossover Bioequivalence Study with a washout period of 7 days. During each session, the subjects were administered a single dose of 100 mg Olaparib Tablets (Test formulation or reference formulation ) under Fasting conditions or 150mg Olaparib Tablets (Test formulation or reference formulation ) under Fasting and Fed conditions. Venous blood samples were collected at pre-dose (0 h), and up to 72 h post dose. This study was to evaluate the bioequivalence and safety of the test formulation and the reference formulation of Olaparib Tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were fully aware of the purpose, character, methodology, and possible adverse effects of the trial, and signed an informed consent form prior to the initiation of any research procedures;
2. Healthy male aged 18 to 50 years old (including critical values);
3. Weight equal to or more than 50.0 kg and body mass index between 19 to 26.0 kg/m^2 (including critical values);
4. Participants had no history of chronic or serious diseases, including cardiovascular, respiratory, gastrointestinal, urinary, hematologic and lymphatic, endocrine, immune, psychiatric, or neurological system diseases;
5. Participants whose immediate family members had no breast, ovarian, pancreatic, prostate cancer, and other related diseases;
6. Normal or abnormal results without clinical significance on all tests including vital signs, physical examination, laboratory evaluation (hematology, urinalysis, blood biochemistry, serology, coagulation function, and urine drug screening), 12-lead electrocardiogram, chest X-ray /Chest Computed Tomography (CCT) and alcohol breath test;
7. Voluntarily signed the informed consent form, and cooperated in completing the trial according to the protocol.

Exclusion Criteria:

1. Allergic constitution or allergic history to drugs or food;
2. Participants with tablet swallowing distress;
3. Participants with a history of surgery or trauma that may affect safety or in vivo metabolism of the drug, or who had undergone surgery within 1 year prior to screening or who were scheduled to undergo surgery during the trial;
4. Participants who had used potent CYP 3A4 strong inhibitors, CYP 3A4 moderate inhibitors, CYP 3A4 strong inducers, and CYP 3A4 moderate inducers within 4 weeks prior to screening;
5. Participants who had used p-gp inhibitors within 4 weeks prior to screening;
6. Participants who had used any medicines or health products within 2 weeks prior to screening,
7. Participants with a history of drug or substance abuse within 6 months prior to screening,or a positive urine drug test during screening;
8. Participants who had used drugs within 3 months prior to screening;
9. Smoking ≥ 5 cigarettes per day on average within 3 months prior to screening,or participants who could not stop using any tobacco-based products during the trial period;
10. Participants who consumed more than 14 units of alcohol per week within the 3 months prior to screening, or who had a positive breath test for alcohol at screening,or who could not abstain from alcohol during the trial ;
11. Participants who consumed excessive amounts of tea, coffee and/or caffeine-rich beverages per day within 3 months prior to screening
12. Participants who had taken a special diet (dragon fruit, mango, grapefruit, lime, star fruit or food or drink prepared from them) within 7 days prior to screening, or participants who were unable to stop taking the above special diets during the trial;
13. Participants who had participated in other clinical trials within 3 months prior to screening;
14. Participants who had lost blood or donated more than 400 ml of blood or who had received blood transfusions or used blood products within 3 months prior to screening;
15. Participants who cannot tolerate venipuncture or with a history of fainting needle or blood;
16. Participants who are lactose intolerant;
17. Participants with special dietary requirements who could not accept a uniform diet;
18. Participants who were planning to have children, unwilling or unable to use effective contraception, or had a plan to donate sperm from 2 weeks prior to the screening until 6 months after the last dose of study drug, and who were unwilling to use non-pharmacological contraception from 2 weeks prior to the screening until one month after the last dose of study drug;
19. Any condition that the investigator considered inappropriate for participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male only
Enrollment: 102 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Cmax Description: Maximum observed plasma concentration | Up to 72 hours post-dose for each period
  Cmax Description: Maximum observed plasma concentration
AUC0-∞ Description: Area under the plasma concentration time curve from time zero extrapolated to infinite time | Up to 72 hours post-dose for each period
  AUC0-∞ Description: Area under the plasma concentration time curve from time zero extrapolated to infinite time
AUC0-t Description: Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration | Up to 72 hours post-dose for each period
  AUC0-t Description: Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 72 hours post-dose for each period
  Time of maximum observed plasma concentration (Tmax)
Terminal elimination half-life (T1/2) | Up to 72 hours post-dose for each period
  Terminal elimination half-life (T1/2)
Apparent total body clearance (Cl/F) | Up to 72 hours post-dose for each period
  Apparent total body clearance (Cl/F)
Apparent volume of distribution (V/F) | Up to 72 hours post-dose for eachperiod
  Apparent volume of distribution (V/F)
Number of participants with Adverse Events | Up to 10 days
  Number of participants with Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China